CLINICAL TRIAL: NCT01182545
Title: A Prospective Randomized Study of the Effects of Hyperventilation Prior to Carbon Dioxide Insufflation on Hemodynamic Changes During Laparoscopic Cholecystectomy
Brief Title: The Effects of Hyperventilation Prior to CO2 Insufflation During Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal University (Other)
Responsible Party: Dr. Mohamed El Tahan, King Faisal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-10-2007
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Anaesthesia; laparoscopic cholecystectomy; CO2 insufflation; hemodynamic; hyperventilation
MeSH Terms: conditions — Hyperventilation | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The normoventilation group (Placebo Comparator): 15 minutes prior to CO2 insufflation, the patients' lungs were ventilated with a tidal volume (TV) of about 8 mL.kg-1 and respiratory rate (R.R) owas adjusted to maintain an end-tidal CO2 (ETCO2) of 4.6-6 kPa throughout the procedure.
  Interventions: Procedure: Ventilation
- The hyperventilation group (Active Comparator): 15 minutes prior to CO2 insufflation, the patients' lungs were ventilated with a TV of 8 mL.kg-1 with the adjustment of the R.R to maintain an ETCO2 of 4-4.6 kPa, until the end of anaesthesia.
  Interventions: Procedure: Ventilation

INTERVENTIONS:
Procedure: Ventilation — Mechanical ventilation was conducted in all the patients with a Datex-Ohmeda Aestiva/5 Smart Ventilator (Madison, WI) through a rebreathing circuit incorporating a CO2 absorber, a heat and moisture exchanger using volume-controlled mode with an inspiratory to expiratory ratio of 1:2.5, and positive end-expiratory pressure (PEEP) of 5 cm H2O. Plateau pressure was kept as low as possible with an upper limit of 30 cm H2O, and the absence of auto-PEEP was ensured by a drop of the expiratory flow to zero on the flow-time curve.

SUMMARY:
The investigators postulated that the use of hyperventilation after induction of anesthesia before CO2 insufflation for laparoscopic surgery in Trendelenburg position would maintain normocapnia and reduce the hemodynamic percussion response of CO2 insufflation.

DETAILED DESCRIPTION:
The use of laparoscopic techniques has become common in clinical practice. Absorption of carbon dioxide (CO2) from the peritoneal cavity is the potential mechanism for hypercapnia and a rise in the end-tidal carbon dioxide (EtCO2). Mild hypercarbia causes sympathetic stimulation which results in a fivefold increase in arginine vasopressin (AVP), tachycardia, increased systemic vascular resistance, systemic arterial pressure, central venous pressure and cardiac output.1 Severe hypercarbia exerts a negative inotropic effect on the heart and reduces left ventricular function.2 Hemodynamic alterations occur only when the PaCO2 is increased by 30 per cent above the normal levels.

Clearance of CO2 is a function of the adequacy of alveolar ventilation with respect to pulmonary perfusion. Controlled hyperventilation has proved to be superior over spontaneous respiration or controlled normo-ventilation for maintaining normal PCO2 during laparoscopy. During pelvic laparoscopy there was a rapid rise of about 30% in the CO2 load eliminated by the lungs. This quickly reached a plateau and could be compensated by hyperventilation of the lungs with a 30% increase in minute ventilation.

Papadimitriou and co' workers concluded that under sevoflurane anesthesia MAC, prophylactic hyperventilation to ensure mild hypocapnia, (around 33 mmHg) limits the cerebral blood flow velocities enhancing effect of CO2 insufflation, compared with permissive hypercapnia (up to 45 mmHg), during gynecological laparoscopies. However, others advocated that hyperventilation and the head-up position before CO2 insufflation are not sufficient to prevent the CO2-mediated cerebral hemodynamic effects of low-pressure pneumoperitoneum (5-8 mmHg) in children, underwent laparoscopic fundoplication.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* aged 18-45 years
* undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* history of cardiovascular disease
* respiratory diseases
* neurological disease
* renal disease
* liver disease
* hormonal disease
* pregnancy
* obesity (defined as a body mass index> 29)
* smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
haemodynamic percussion response | at 5 and 10 minutes, in supine and Trendelenburg (30° head-down) positions, respectively, before CO2 insufflation and at 15, 30, 45, and 60 min after CO2 insufflation, and at 5 min after desufflation of pneumoperitoneum
  changes in mean arterial blood pressure [MAP] and heart rate [H.R].

SECONDARY OUTCOMES:
other hemodynamic and respiratory parameters | at 5 and 10 minutes, in supine and Trendelenburg (30° head-down) positions, respectively, before CO2 insufflation and at 15, 30, 45, and 60 min after CO2 insufflation, and at 5 min after desufflation of pneumoperitoneum,
  systemic vascular resistance index (SVRI), cardiac index (CI), stroke volume index (SVI), PaCO2, EtCO2, arterial to end-tidal CO2 gradient (Pa-EtCO2), respiratory rate and airway pressures were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D., Study Director — King Faisal University
Locations (1):
- King Faisal University, Khobar, Eastern Province, Saudi Arabia